CLINICAL TRIAL: NCT01370161
Title: Early Transjugular Intrahepatic Portosystemic Shunt With Polytetrafluoroethylene Covered Stents Versus Standard Medical Therapy for Acute Variceal Bleeding in Patients With Advanced Cirrhosis
Brief Title: Early TIPS With Polytetrafluoroethylene (PTFE) Covered Stents for Acute Variceal Bleeding in Patients With Advanced Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHDD 002; FMMU-XHDD 002 (Registry Identifier: Fourth Military Medical University)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Decompensated Cirrhosis; Bleeding Varices
Keywords: transjugular intrahepatic portosystemic shunt; TIPS; variceal bleeding; liver cirrhosis; hepatitis B
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B | interventions — Portasystemic Shunt, Transjugular Intrahepatic

ARMS (2):
- TIPS treatment (Experimental): Initial control of the bleeding episode will be obtained by vasoactive drugs (octreotide, somatostatin or terlipressin), endoscopic band ligation (sclerotherapy if technically difficult or not feasible) and prophylactic antibiotics.TIPS will be performed as soon as possible once the patients are enrolled in the study, always within the first 72 hours after the diagnostic endoscopy (preferably in the first 24 hours).Vasoactive drugs will be continued until the TIPS is performed and antibiotics will be continued for 5-7 days.
  Interventions: Procedure: TIPS treatment
- Medical treatment (Active Comparator): Initial control of the bleeding episode will be obtained by vasoactive drugs (octreotide, somatostatin or terlipressin), endoscopic band ligation (sclerotherapy if technically difficult or not feasible) and prophylactic antibiotics.Patients will be treated with non-selective beta-blockers (propranolol)on day 5. In case of contraindications or intolerance to beta-blockers, patients will not receive pharmacological treatment (beta-blockers) and the only treatment to prevent rebleeding will be endoscopic band ligation.
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Procedure: TIPS treatment — 1. A 8 mm Fluency stent will be used. The aim will be to reduce the portal pressure gradient (PPG) below to 12 mm Hg or 25-75% of baseline.
  2. Embolisation, either with coils or bucrylate, can be performed, if it is felt necessary, especially in patients where portography shows the filling of large portosystemic collaterals feeding the varices.
  3. After TIPS, anticoagulation will not be used as a rule, but is allowed if the attending physician thinks that it is warranted.
  Other Names: Transjugular intrahepatic portosystemic shunt (TIPS)
  Arms: TIPS treatment
Drug: Medical treatment — Patients will receive vasoactive drugs up to 5 days; then a non-selective beta-blocker (propranolol) will be started with an initial dose of 40 mg, the dose of propranolol will be increased/decreased step by step to achieve a baseline heart rate of 55 bpm, or 25% reduction of basal heart rate or up to the maximum tolerated dose of propranolol.
  The second elective session of endoscopic band ligation will be performed within the first 7-14 days after the initial endoscopic treatment. The following sessions will be performed at 14 +/- 3 days intervals until variceal eradication. Once eradication is achieved, endoscopic monitoring will be performed every 6 months. If varices reappear, new band ligation will be performed.
  Other Names: Non-selective beta blocker + Endoscopic variceal ligation
  Arms: Medical treatment

SUMMARY:
The purpose of this study is to determine whether early use of transjugular intrahepatic portosystemic shunt (TIPS) with Polytetrafluoroethylene (PTFE) covered stents is able to prolong the survival in patients with advanced cirrhosis and acute variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* History of cirrhosis (clinical or by liver biopsy)
* Admission due to acute bleeding from oesophageal or gastric (GOV1 or GOV2) varices
* Child-Pugh Class C (Child-Pugh score less than or equal to 13) or Child-Pugh class B
* Signed written informed consent

Exclusion Criteria:

* Patients not fulfilling inclusion criteria
* Pregnancy or breast-feeding
* Confirmed hepatocellular carcinoma
* Creatinine greater than 3 mg/dl
* Terminal hepatic failure (Child-Pugh score greater than 13)
* Previous treatment with TIPS or combined pharmacological and endoscopic treatment to prevent rebleeding
* Fundal or ectopic gastric variceal bleeding (IGV1 or IGV2)
* Complete portal vein thrombosis or portal cavernoma
* Congestive heart failure New York Heart Association (NYHA) greater than III or medical history of pulmonary hypertension
* Spontaneous recurrent hepatic encephalopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-07; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of survival without liver transplantation | 2 years

SECONDARY OUTCOMES:
Number of participants failed to control acute variceal bleeding within 5 days, 6 weeks and 1 year | 1 years
Number of bleeding related death | 2 years
Number of other portal hypertension related complications on follow-up (ascites, hepatorenal syndrome, hepatic encephalopathy) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD & MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Garcia-Pagan JC, Caca K, Bureau C, Laleman W, Appenrodt B, Luca A, Abraldes JG, Nevens F, Vinel JP, Mossner J, Bosch J; Early TIPS (Transjugular Intrahepatic Portosystemic Shunt) Cooperative Study Group. Early use of TIPS in patients with cirrhosis and variceal bleeding. N Engl J Med. 2010 Jun 24;362(25):2370-9. doi: 10.1056/NEJMoa0910102. PMID 20573925
- [Derived] Lv Y, Yang Z, Liu L, Li K, He C, Wang Z, Bai W, Guo W, Yu T, Yuan X, Zhang H, Xie H, Yao L, Wang J, Li T, Wang Q, Chen H, Wang E, Xia D, Luo B, Li X, Yuan J, Han N, Zhu Y, Niu J, Cai H, Xia J, Yin Z, Wu K, Fan D, Han G; AVB-TIPS Study Group. Early TIPS with covered stents versus standard treatment for acute variceal bleeding in patients with advanced cirrhosis: a randomised controlled trial. Lancet Gastroenterol Hepatol. 2019 Aug;4(8):587-598. doi: 10.1016/S2468-1253(19)30090-1. Epub 2019 May 29. PMID 31153882